CLINICAL TRIAL: NCT04319380
Title: Seasonal Vaccination With the RTS,S/AS01 Malaria Vaccine Given With or Without Seasonal Malaria Chemoprevention: Extension of a Randomised, Double-blind Phase 3 Trial Until Children Reach the Age of Five Years
Brief Title: Seasonal Malaria Vaccination (RTS,S/AS01) and Seasonal Malaria Chemoprevention (SP/AQ) Extension Study
Acronym: RTSS-SMC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RTS,S + SMC extn
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-01

CONDITIONS: Malaria,Falciparum; Child, Only
Keywords: Malaria; Seasonal vaccination; Seasonal chemoprevention
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Tetanus Toxoid; Clinical Trials Data Monitoring Committees; RTS,S-AS01 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMC with SP+AQ (Active Comparator): Administration of tetanus/diphtheria toxoids vaccine followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1 and 2.
  Interventions: Biological: Tetanus/diphtheria toxoids; Drug: SMC with SP+AQ
- RTS,S/AS01 (Active Comparator): Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with placebo in Year 1 and 2.
  Interventions: Biological: RTS,S/AS01; Drug: SMC placebo
- RTS,S/AS01 plus SMC with SP+AQ (Active Comparator): Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1 and 2.
  Interventions: Drug: SMC with SP+AQ; Biological: RTS,S/AS01

INTERVENTIONS:
Biological: Tetanus/diphtheria toxoids — One dose of tetanus/diphtheria toxoids vaccine (June) in year 1 and year 2.
  Arms: SMC with SP+AQ
Drug: SMC with SP+AQ — Year 1 and 2 (2020/21) Four cycles of SMC (SP+AQ) (July, August, September, October). One cycle of SMC consisting of sulphadoxine - pyrimethamine (SP) 500mg/25 mg, and amodiaquine (AQ) 150mg on day 1, and AQ 150mg on days 2 and 3.
  Arms: RTS,S/AS01 plus SMC with SP+AQ; SMC with SP+AQ
Biological: RTS,S/AS01 — One booster dose of RTSS/AS01 (June) in year 1 and 2.
  Arms: RTS,S/AS01; RTS,S/AS01 plus SMC with SP+AQ
Drug: SMC placebo — Year 1 and 2 (2020/21) Four cycles of SMC placebo (July, August, September, October)
  Arms: RTS,S/AS01

SUMMARY:
A double-blind, individual randomised trial will be undertaken in children under five years of age living in areas of Burkina Faso or Mali where the transmission of malaria is intense and highly seasonal to determine whether administration of further doses of the malaria vaccine RTS,S/AS01 at the beginning of the malaria transmission until children reach the age of five years is (a) as effective as SMC with SP + AQ in preventing clinical malaria (b) provides additional, useful protection when given together with SMC. The primary trial end-point will be the incidence of clinical episodes of malaria detected by passive case detection. This is a two year extension of the current RTS,S/AS01 + SMC trial to continue the trial until the study children reach the age of five years, the current age at which SMC is recommended until.

DETAILED DESCRIPTION:
Although there has been substantial progress in malaria control in the past decade, this progress has stalled in many countries in sub-Saharan Africa, especially in countries of the Sahel and central Africa, despite widespread deployment of insecticide treated bednets, chemoprevention and improved access to treatment. Recognition of this new challenge has led WHO's Global Malaria Programme (GMP) to establish a new 'High Burden, High Impact' programme which focuses on 10 countries in Africa, including Burkina Faso and Mali, and India. In these countries, where current control and treatment measure are failing to bring malaria fully under control, new approaches to malaria control are needed.

The RTS,S/AS01 malaria vaccine is a recombinant protein vaccine in which the fusion protein RTS (containing parts of the circumsporozoite protein (CSP) of Plasmodium falciparum fused to hepatitis B surface antigen (HBsAg)) is co-expressed in yeast together with free HBsAg (S) to form a virus like particle (RTS,S); it is given with the powerful adjuvant AS01. RTS,S/AS01 induces a strong antibody response to the P. falciparum CSP and high titres of anti-CSP antibody are associated with protection. Following a long process of development, a phase 3 study of RTS,S/AS01 conducted in 15,439 children in 7 countries in Africa showed that three doses of RTS,S/AS01 given with a one month interval between doses, followed by a fourth dose 18 months post dose 3, gave 36.5 % [95% CI 31,41%] protection against clinical attacks of malaria when given to young children aged 5-17 months who were followed for 48 months; efficacy was less when given to infants at the age of 6-12 weeks. RTS,S/AS01 provides a high level of protection during the first three months after vaccination, modelled to be about 70% in the phase 3 trial, a level of initial efficacy similar to that observed in an earlier phase 2 trial in Gambian adults. However, efficacy wanes progressively over the following months. A subsequent dose given 18 months after the primary series restores some but not all of the efficacy seen immediately after the primary series. In July 2015, the European Medicines Agency reviewed efficacy and safety data on RTS.S/AS01 and concluded that the risk benefit balance favoured the vaccine and gave a positive opinion on its use in children aged 6 weeks to 17 months. One potential use for the RTS,S/AS01 vaccine is to use it to prevent seasonal malaria, taking advantage of its high but rapidly waning efficacy.

Across the African Sahel and sub-Sahel, where malaria transmission is very high and concentrated in a few months of the year, Seasonal Malaria Chemoprevention (SMC),a malaria control intervention in which children under the age of five years, the group most at risk, are given the antimalarials sulphadoxine pyrimethamine and amodiaquine (SP+AQ) at monthly intervals for four months during the peak malaria transmission season, has proved very effective. However, the delivery of SMC is demanding on the recipient and provider, requiring four contacts each malaria transmission season if anti-malarials are given to mothers to administer at home and 12 contacts if directly observed treatment is employed. In addition, SMC is threatened by the emergence of resistance to SP and AQ and there are currently no other combinations of licensed antimalarials that could be used to replace them. It is likely to be 5-10 years before novel antimalarials under development could be deployed for SMC. In contrast to SMC, seasonal vaccination with RTS,S/AS01 would require only one visit each transmission season after priming. RTS,S/AS01 may be a little less effective than SMC during the malaria transmission season but this may be balanced by provision of protection during the dry season, when some malaria transmission still occurs and when SMC would provide no benefit. There is, therefore, a need for a comparative study of these two interventions. In some areas where SMC is currently being deployed, and other malaria control interventions such as long-lasting insecticide treated nets used widely, the incidence of malaria in young children remains high (0.4 episodes per year in children under the age of five years in SMC recipients in Burkina Faso). Thus, determining whether RTS,S/AS01 would provide added, useful protection to SMC in such situations is also important. It might also be able to protect some children who, because of side effects, are unable or unwilling to take SMC.

Thus, in 2017, a double-blind, individual randomised trial trial was started in Mali and Burkina Faso to investigate the beneficial effects of adding the RTS,S/AS01 malaria vaccine to SMC and to determine whether it might be possible to replace SMC with RTS,S/AS01. The RTS,S/AS01 + SMC trial, which is supported by the UK Global Clinical Trials Programme and PATH, recruited 5887 children aged 5-17 months in Burkina Faso and Mali who have been randomised to one of three trial groups (a) SMC + RTS,S/AS01 (b) RTS,S/AS01 + a SMC placebo or (c) SMC + a control vaccine. Study children have now been followed through three malaria transmission seasons and the first phase of the trial will finish in April 2020. This trial will now be extended for two years until the study children reach the age of five years, the current age at which SMC is recommended until.

ELIGIBILITY:
Inclusion Criteria:

* The child had been enrolled in the initial phase of the trial of seasonal vaccination with the RTS,S/AS01 vaccine
* A parent or legally recognised guardian provides informed consent for the child's inclusion in the extension study
* The child is a permanent resident of the study area and likely to remain a resident for the duration of the trial

The child is under five years of age at the time of enrolment.

Exclusion Criteria:

* The child has had an allergic reaction to the study drugs or vaccines
* The child had febrile convulsions on more than one occasion following vaccination
* The child has developed a serious underlying illness such as severe malnutrition (weight for age or mid arm circumference Z scores < 3 SD) which in view of the investigators might impair the response to vaccination
* The child has been enrolled in another malaria vaccine or other experimental malaria intervention study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5098 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, Professor, Study Director — Malaria Research & Training Center, Bamako; Jean Bosco Ouedraogo, Professor, Study Director — Institut de Recherche en Sciences de la Santé, Direction Régionale de l'Ouest (IRSS-DRO)
Locations (2):
- Institut de Recherche en Sciences de la Santé, Ouagadougou, Direction Régionale de l'Ouest, Burkina Faso
- Malaria Research & Training Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the LSHTM Data Compass system

REFERENCES:
- [Derived] Dicko A, Ouedraogo JB, Zongo I, Sagara I, Cairns M, Yerbanga RS, Issiaka D, Zoungrana C, Sidibe Y, Tapily A, Nikiema F, Sompougdou F, Sanogo K, Kaya M, Yalcouye H, Dicko OM, Diarra M, Diarra K, Thera I, Haro A, Sienou AA, Traore S, Mahamar A, Dolo A, Kuepfer I, Snell P, Grant J, Webster J, Milligan P, Lee C, Ockenhouse C, Ofori-Anyinam O, Tinto H, Djimde A, Chandramohan D, Greenwood B. Seasonal vaccination with RTS,S/AS01E vaccine with or without seasonal malaria chemoprevention in children up to the age of 5 years in Burkina Faso and Mali: a double-blind, randomised, controlled, phase 3 trial. Lancet Infect Dis. 2024 Jan;24(1):75-86. doi: 10.1016/S1473-3099(23)00368-7. Epub 2023 Aug 22. PMID 37625434

RESULTS

PARTICIPANT FLOW:
Groups:
- SMC With SP+AQ: Administration of tetanus/diphtheria toxoids vaccine followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1 and 2.
  Tetanus/diphtheria toxoids: One dose of tetanus/diphtheria toxoids vaccine (June) in year 1 and year 2.
  SMC with SP+AQ: Year 1 and 2 (2020/21) Four cycles of SMC (SP+AQ) (July, August, September, October). One cycle of SMC consisting of sulphadoxine - pyrimethamine (SP) 500mg/25 mg, and amodiaquine (AQ) 150mg on day 1, and AQ 150mg on days 2 and 3. In Year 2 (2021), a fifth cycle of SMC with SP+AQ was given to children in Burkina Faso in line with national guidelines.
- RTS,S/AS01: Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with placebo in Year 1 and 2.
  RTS,S/AS01: One booster dose of RTSS/AS01 (June) in year 1 and 2.
  SMC placebo: Year 1 and 2 (2020/21) Four cycles of SMC placebo (July, August, September, October). In Year 2 (2021), a fifth cycle of SMC placebo was given to children in Burkina Faso in line with national guidelines.
- RTS,S/AS01 Plus SMC With SP+AQ: Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1 and 2.
  SMC with SP+AQ: Year 1 and 2 (2020/21) Four cycles of SMC (SP+AQ) (July, August, September, October). One cycle of SMC consisting of sulphadoxine - pyrimethamine (SP) 500mg/25 mg, and amodiaquine (AQ) 150mg on day 1, and AQ 150mg on days 2 and 3. In Year 2 (2021), a fifth cycle of SMC with SP+AQ was given to children in Burkina Faso in line with national guidelines.
  RTS,S/AS01: One booster dose of RTSS/AS01 (June) in year 1 and 2.
Period: Overall Study
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 Plus SMC With SP+AQ
Started | 1683 | 1705 | 1710
Completed | 1644 | 1650 | 1661
Not Completed | 39 | 55 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 Plus SMC With SP+AQ | Total
Number analyzed (Participants) | 1683 | 1705 | 1710 | 5098
Age, Continuous [Mean (Standard Deviation); unit: Months] | 48.6 (4.3) | 48.8 (4.2) | 48.6 (4.2) | 48.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 817 | 813 | 830 | 2460
  Male | 866 | 892 | 880 | 2638
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 824 | 813 | 837 | 2474
  Mali | 859 | 892 | 873 | 2624

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Episodes of Malaria
Description: Passive surveillance to detect episode of fever (temperature > 37.5 C), or a history of fever within the past 48 hours, that is severe enough to require treatment at a health centre and which is accompanied by a positive blood film with a parasite density of 5,000 per µl or more
Time Frame: Passive surveillance of clinical episodes of malaria within the study area over 24 months (1 April 2020 until 31 March 2022).
Measure: Number (95% Confidence Interval); unit: Episodes per 1,000 child years at risk
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 Plus SMC With SP+AQ
Number analyzed (Participants) | 1683 | 1705 | 1710
Episodes per 1,000 child years at risk | 338.1 [315.4 to 362.2] | 421.3 [395.5 to 448.2] | 178.9 [162.5 to 196.7]

2. Secondary Outcome: Clinical Episodes of Uncomplicated Febrile Illness
Description: Passive and active surveillance to detect cases with temperature > 37.5o C), or a history of fever within the past 48 hours, with a positive blood film (any level of asexual parasitaemia) or a positive rapid diagnostic test (RDT) for malaria
Time Frame: Passive surveillance in all health centers within the study area starting 1 April 2020 until 31 March 2022.
Reporting Status: Not Posted

3. Secondary Outcome: Hospital Admissions With Malaria, Including Severe Malaria
Description: Hospital admissions with malaria, including cases of severe malaria which meet WHO criteria for a diagnosis of severe malaria.
Time Frame: Through study completion, each child admitted in a study hospital will be treated and monitored until complete cure or death (a period of 2 years). Documentation of each hospital admission according to ICH-GCP
Reporting Status: Not Posted

4. Secondary Outcome: Prevalence of Malaria Parasitaemia, Including Gametocytaemia and the Prevalence of Moderate and Severe Anemia and Malnutrition
Description: The prevalence of malaria parasitaemia, including gametocytaemia, moderate and severe anaemia and malnutrition at the end of the malaria transmission season
Time Frame: Blood sample collection during 2-week cross sectional survey at the end of each malaria transmission season (November 2020/21).).
Reporting Status: Not Posted

5. Secondary Outcome: Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs), including any deaths, occurring at any time during the study with special reference to any cases of meningitis and cerebral malaria (WHO case definition)
Time Frame: Through study completion (for 2 years), each SAE will be treated and documented according to ICH-GCP.
Reporting Status: Not Posted

6. Secondary Outcome: Immune Response to the Vaccine (Anti-CSP Antibody Concentrations)
Description: Anti-CSP antibody concentrations obtained before and after each booster dose, determined in a sub-sample of children.
Time Frame: Blood sample collection 0-7 days before and one month after the booster doses (year 1 and 2).
Reporting Status: Not Posted

7. Secondary Outcome: Prevalence of Malaria Parasitaemia in School Aged Children
Description: The prevalence of malaria parasitaemia at the end of each malaria transmission season in school-age children resident in the study areas, to determine overall malaria transmission
Time Frame: Blood sample collection during the 2-week cross sectional survey at the end of each malaria transmission season (November 2020/21).
Reporting Status: Not Posted

8. Secondary Outcome: Polymorphisms in the P. Falciparum CSP
Description: The prevalence of mutations in the Th2 or Th3 locus of the Plasmodium falciparum csp gene in isolates from children who have received RTS,S/AS01 that differ from those of the isolate used in the preparation of the vaccine
Time Frame: Blood sample collection from children with clinical episodes of malaria and in children with parasitaemia at the 2-week cross-sectional survey (November 2020/21)).
Reporting Status: Not Posted

9. Secondary Outcome: Drug Resistance to SP and AQ
Description: The presence of molecular markers of resistance to SP and AQ in parasite positive samples
Time Frame: Blood sample collection during the final 2-week cross sectional survey conducted at the end of malaria transmission season (November 2021)
Reporting Status: Not Posted

10. Secondary Outcome: SP+AQ Drug Sensitivity
Description: The 28-day treatment outcome in children with asymptomatic malaria parasitaemia treated with SP+AQ.
Time Frame: Children with asymptomatic malaria parasitaemia identified during the final cross-sectional survey (November 2021), treated with a full course of SP+AQ over 3 days and followed for 28 days.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious adverse event data were collected over a 24 month period (1st April 2020 to 31st March 2022).
Description: The number of participants at risk for other (non-serious) adverse events is zero because non-serious adverse events were not collected or assessed as part of this study.
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 Plus SMC With SP+AQ
All-Cause Mortality (participants affected / at risk) | 2/1683 | 10/1705 | 4/1710
Serious Adverse Events (participants affected / at risk) | 11/1683 | 16/1705 | 16/1710
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMC With SP+AQ (N=1683) | RTS,S/AS01 (N=1705) | RTS,S/AS01 Plus SMC With SP+AQ (N=1710)
Hospitalisations (all causes) (General disorders) | 11 | 16 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04319380/Prot_SAP_000.pdf